CLINICAL TRIAL: NCT07089368
Title: Photodynamic Therapy With Topical Application of a Zn(II) Phthalocyanine (RLP068/Cl) and Red Light for the Treatment of Moderate-to-severe Acne Vulgaris
Acronym: PHOTAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Stefano Bighetti, MD, Università degli Studi di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025BSDR09C
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-04

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RLP068/Cl Photodynamic Therapy (Experimental)
  Interventions: Drug: Zn(II)-phthalocyanine gel

INTERVENTIONS:
Drug: Zn(II)-phthalocyanine gel — Topical application of RLP068/Cl 0.3% gel (Zn(II)-phthalocyanine) at a dose of 1 mL per 25 cm² under occlusion for 30 minutes, followed by red light irradiation at 630 nm (60 J/cm²) for 8 minutes. Sessions will be repeated twice weekly until clinical response is achieved.

SUMMARY:
This pilot clinical study will evaluate the safety, tolerability, and effectiveness of a novel photodynamic therapy (PDT) for moderate-to-severe acne vulgaris. PDT combines a topical photosensitizing gel with red light to treat acne lesions. The gel to be used in this study, called RLP068/Cl (a zinc phthalocyanine compound), has demonstrated antimicrobial, anti-inflammatory, and sebosuppressive effects in laboratory studies.

A total of 10 patients with moderate-to-severe acne on the face will be enrolled. RLP068/Cl 0.3% gel will be applied topically for 30 minutes under occlusion, followed by 8 minutes of red LED light exposure. Treatments will be performed twice weekly, with the total number of sessions individualized based on clinical response.

Acne severity will be assessed using the Global Acne Grading System (GAGS). Pain levels will be recorded after each session using a visual scale, and patient satisfaction will be evaluated at the end of the treatment cycle.

The goal of the study is to determine whether RLP068/Cl-PDT is a safe, well-tolerated, and effective non-antibiotic treatment option for patients with moderate-to-severe acne vulgaris who may not respond to or tolerate conventional therapies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged ≥16 years.
* Diagnosis of moderate-to-severe acne vulgaris (comedonal, papulopustular, or cystic), with facial lesions symmetrically distributed.
* Washout period of at least 6 months from prior oral acne treatments.
* Washout period of at least 2 months from prior topical acne treatments.
* Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

* Use of systemic or topical photosensitizing medications.
* Known photosensitivity disorders.
* Pregnancy or breastfeeding.
* Participation in another interventional clinical study within the past 3 months.
* Any dermatological condition of the face that may interfere with treatment assessment (e.g., eczema, rosacea).
* Any serious uncontrolled medical condition deemed by the investigator to pose a risk to the participant or interfere with study results.

Min Age: 16 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Global Acne Grading System (GAGS) score from baseline | End of treatment (EOT), expected within 4 to 6 weeks from baseline
  The Global Acne Grading System (GAGS) is a validated tool that assesses acne severity based on lesion type and anatomical location. The outcome will be measured as the change in total GAGS score from baseline to the end of treatment.

IPD SHARING:
Plan to Share IPD: Yes